CLINICAL TRIAL: NCT00003864
Title: A Phase II Trial of Docetaxel and Carboplatin in Patients With Advanced Squamous Carcinoma of the Esophagus
Brief Title: Docetaxel Plus Carboplatin in Treating Patients With Advanced Cancer of the Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067028; E-2298
Record Dates: First submitted 1999-11-01; First posted 2004-04-02 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Cancer
Keywords: stage III esophageal cancer; stage IV esophageal cancer; squamous cell carcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Carboplatin; Docetaxel

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of docetaxel plus carboplatin in treating patients who have advanced cancer of the esophagus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the objective response rate in patients with advanced squamous cell carcinoma of the esophagus treated with carboplatin and docetaxel. II. Assess the toxicity of this regimen in these patients. III. Assess the time to progression and overall survival of this patient population.

OUTLINE: Patients receive docetaxel IV over 1 hour on day 1, followed by carboplatin IV over 15-30 minutes on day 1. Treatment is repeated every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months until year 2, every 6 months during years 2-5, and then annually thereafter until death.

PROJECTED ACCRUAL: A total of 18-35 patients will be accrued for this study at a rate of 30 patients per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic or incurable, locally advanced squamous cell carcinoma of the esophagus Measurable disease outside of a previously radiated field required

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal SGOT no greater than 2 times upper limit of normal Renal: Creatinine normal Cardiovascular: No congestive heart failure or angina pectoris, even if medically controlled No prior myocardial infarction within the past year No clinically significant conduction system abnormalities, such as 2nd or 3rd degree heart block or bundle branch block Pulmonary: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception No active infections or medical illnesses that are uncontrolled No second malignancy other than previously treated nonmelanoma skin cancer or carcinoma in situ of the cervix or a prior malignancy from which patient has been disease free for past 3 years Caloric intake greater than 1500 calories/day Fluid intake greater than 1500 mL/day

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09-03 (Actual); Primary Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coenraad F. Slabber, MD, Study Chair — Pretoria Academic Hospital
Locations (74):
- United States (71):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Cancer Center and Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Raritan Bay Medical Center, Perth Amboy, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Result] Rossman JF, Falkson CI, Xu R, Slabber CF, Mason BA, Mulcahy MF, Benson AB 3rd. Phase II Trial of Docetaxel and Carboplatin in Patients With Advanced Squamous Carcinoma of the Esophagus (E2298): A Trial of the Eastern Cooperative Oncology Group. Gastrointest Cancer Res. 2011 Jan;4(1):9-14. PMID 21464865